CLINICAL TRIAL: NCT06826651
Title: Thermal Sealing by Bipolar Diathermy Versus Clips Closure of Mesoappendix in Laparoscopic Appendectomy ..A Comparative Study
Brief Title: Use of Bipolar Diathermy VS Clips in Laparoscopic Appendectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdulrahman Samir Fahmy Sayed, Resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Use of bipolar diathermy
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Laparoscopic Appendectomy; Bipolar Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Laparoscopic appendectomy, using of bipolar diathermy to coagulate mesoappendix
  Interventions: Procedure: laparoscopic appendectomy; Procedure: bipolar diathermy
- Group B (Experimental): laparoscopic appendectomy, using surgical clips in closure of mesoappendix
  Interventions: Procedure: laparoscopic appendectomy; Procedure: clips closure

INTERVENTIONS:
Procedure: laparoscopic appendectomy — By using laparoscopy, after achieving conclusive identification of the mesoappendix
Procedure: bipolar diathermy — the mesoappendix coagulated using bipolar diathermy, then cut with scissor.
  Arms: Group A
Procedure: clips closure — mesoappendix will be divided between 3 clips, two placed distally and one proximally. The mesoappendix will be cut in between the clips.
  Arms: Group B

SUMMARY:
Acute Appendicitis is the most frequent acute pathological abdominal illness needing immediate surgery. The laparoscopic appendectomy (LA) has become more popular and is advised as the first course of treatment, particularly for female, obese, and elderly patients.LA can also give surgeons a greater field view and identification of other abdominal organs that can have different pathologies that could mimic the symptoms of acute appendicitis.The most crucial step in preventing major complications such postoperative bleeding, peritonitis, sepsis is sealing the mesoappendix. Due to this circumstance, surgeons are looking for alternative treatments for LA. The best technique for sealing mesoappendix should be affordable, practical, safe, and easy to apply technically. Extracorporeal sliding knots, intracorporeal ligations, endo-loops, nonabsorbable polymer clips (Hem-o-lock clips), hand-made loops, and Ligasure usage, and bipolar cautery division are some of the techniques utilized at LA to seal mesoappendix. According to studies, each of these techniques is secure and practicable.5 In this study, there is a comparative study between using Bipolar diathermy as a source of sealing and other mechanical closure techniques for mesoappendix To assess effect of energy source sealing of mesoappendix by using Bipolar diathermy in comparison to mechanical closure by clips as regard outcome and complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to AUH with uncomplicated acute appendicitis or chronic appendicitis
* Age group (18-70)

Exclusion Criteria:

* patients with complex appendicitis (appendicular mass, abscess, etc).
* patients who had the following conditions: cirrhosis with ascites, abdominal distention, and coagulation disorders, cardiac patients; shock upon arrival, a large ventral hernia, and inflammatory bowel disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
intraoperative blood loss | baseline
  amount of blood loss will be calcculated by number of towel used and aomunt of blood in sution